CLINICAL TRIAL: NCT02728492
Title: Open-label Multicenter Multiple Ascending Dose Study to Evaluate Safety, Tolerability and Pharmacokinetics of Quisinostat, a Histone Deacetylase Inhibitor, in Combination With Gemcitabine + Cisplatin Chemotherapy (Second Line for Patients With Non-small Cell Lung Cancer) or Paclitaxel + Carboplatin Chemotherapy (Second Line for Patients With Non-small-cell Lung Cancer, Second and Subsequent Lines for Patients With Epithelial Ovarian Cancer)
Brief Title: Safety, Tolerability and Pharmacokinetics of Quisinostat, a Histone Deacetylase Inhibitor, in Combination With Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewVac LLC (Industry)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-13-NSCLC/OVA-7-QUI-1B
Record Dates: First submitted 2015-11-13; First posted 2016-04-05 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Non-small Cell Lung Cancer; Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial | interventions — quisinostat; Paclitaxel; Carboplatin; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Quisinostat 8 mg & Paclitaxel & Carboplatin (Experimental): Quisinostat 8 mg capsule every other day and Paclitaxel 175 mg/m2 on Day 7 of every 3-weeks course and Carboplatin (mg/ml х min) х [GFR (ml/min) + 25] on Day 7 of every 3-weeks course up to 6 cycles
  Interventions: Drug: Quisinostat; Drug: Paclitaxel; Drug: Carboplatin
- Quisinostat 10 mg & Paclitaxel & Carboplatin (Experimental): Quisinostat 10 mg capsule every other day and Paclitaxel 175 mg/m2 on Day 7 of every 3-weeks course and Carboplatin (mg/ml х min) х [GFR (ml/min) + 25] on Day 7 of every 3-weeks course up to 6 cycles
  Interventions: Drug: Quisinostat; Drug: Paclitaxel; Drug: Carboplatin
- Quisinostat 12 mg & Paclitaxel & Carboplatin (Experimental): Quisinostat 12 mg capsule every other day and Paclitaxel 175 mg/m2 on Day 7 of every 3-weeks course and Carboplatin (mg/ml х min) х [GFR (ml/min) + 25] on Day 7 of every 3-weeks course up to 6 cycles
  Interventions: Drug: Quisinostat; Drug: Paclitaxel; Drug: Carboplatin
- Quisinostat 8 mg & Gemcitabine 1000 mg/m2 & Cisplatin (Experimental): Quisinostat 8 mg capsule every other day and Gemcitabine 1000 mg/m2 on Day 7 and on Day 14 of every 3-weeks course and Cisplatin 75 mg/m2 on Day 7 of every 3-weeks course up to 6 cycles
  Interventions: Drug: Quisinostat; Drug: Gemcitabine; Drug: Cisplatin
- Quisinostat 10 mg & Gemcitabine 1000 mg/m2 & Cisplatin (Experimental): Quisinostat 10 mg capsule every other day and Gemcitabine 1000 mg/m2 on Day 7 and on Day 14 of every 3-weeks course and Cisplatin 75 mg/m2 on Day 7 of every 3-weeks course up to 6 cycles
  Interventions: Drug: Quisinostat; Drug: Gemcitabine; Drug: Cisplatin
- Quisinostat 12 mg & Gemcitabine 1000 mg/m2 & Cisplatin (Experimental): Quisinostat 12 mg capsule every other day and Gemcitabine 1000 mg/m2 on Day 7 and on Day 14 of every 3-weeks course and Cisplatin 75 mg/m2 on Day 7 of every 3-weeks course up to 6 cycles
  Interventions: Drug: Quisinostat; Drug: Gemcitabine; Drug: Cisplatin
- Quisinostat 12 mg & Gemcitabine 1250 mg/m2 & Cisplatin (Experimental): Quisinostat 12 mg capsule every other day and Gemcitabine 1250 mg/m2 on Day 7 and on Day 14 of every 3-weeks course and Cisplatin 75 mg/m2 on Day 7 of every 3-weeks course up to 6 cycles
  Interventions: Drug: Quisinostat; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Quisinostat
  Other Names: JNJ-26481585
Drug: Paclitaxel
  Arms: Quisinostat 10 mg & Paclitaxel & Carboplatin; Quisinostat 12 mg & Paclitaxel & Carboplatin; Quisinostat 8 mg & Paclitaxel & Carboplatin
Drug: Carboplatin
  Arms: Quisinostat 10 mg & Paclitaxel & Carboplatin; Quisinostat 12 mg & Paclitaxel & Carboplatin; Quisinostat 8 mg & Paclitaxel & Carboplatin
Drug: Gemcitabine
  Arms: Quisinostat 10 mg & Gemcitabine 1000 mg/m2 & Cisplatin; Quisinostat 12 mg & Gemcitabine 1000 mg/m2 & Cisplatin; Quisinostat 12 mg & Gemcitabine 1250 mg/m2 & Cisplatin; Quisinostat 8 mg & Gemcitabine 1000 mg/m2 & Cisplatin
Drug: Cisplatin
  Arms: Quisinostat 10 mg & Gemcitabine 1000 mg/m2 & Cisplatin; Quisinostat 12 mg & Gemcitabine 1000 mg/m2 & Cisplatin; Quisinostat 12 mg & Gemcitabine 1250 mg/m2 & Cisplatin; Quisinostat 8 mg & Gemcitabine 1000 mg/m2 & Cisplatin

SUMMARY:
Quisinostat besides its own efficacy, which can potentially lead to better results of polychemotherapy and increase the mean time to progression, it may be demonstrated that Quisinostat leads to sustained tumor sensitivity to platinum drugs. In this study safety and tolerability of multiple administrations of Quisinostat in doses ranging from 8 mg to 12 mg combined with standard backbone chemotherapy in patients with non-small cell lung cancer (second line) and ovarian cancer (second and subsequent lines) will be investigated.

DETAILED DESCRIPTION:
It was proven that Quisinostat increases HDAC1-inhibited E-cadherin expression (at the low concentrations of 30 nM) which increases susceptibility to epidermal growth factor inhibitors in case of non-small-cell lung cancer and stops proliferation of paclitaxel-resistant cells. Thus, besides its own efficacy, which can potentially lead to better results of polychemotherapy and increase the mean time to progression, it may be demonstrated that Quisinostat leads to sustained tumor sensitivity to platinum drugs and possibly to resensitiztion in case of acquired or primary resistance.

The main objective of the study is to evaluate the safety and tolerability of Quisinostat in multiple ascending doses and establish its maximum tolerated dose (MTD), administered in combination with standard backbone chemotherapy, as follows: Gemcitabine + Cisplatin in patients with non-small-cell lung cancer (second line) and Paclitaxel + Carboplatin in patients with non-small-cell lung cancer (second line) and in patients with ovarian cancer (second and subsequent lines). MTD is defined as maximum dose at which DLT occurs in no more than 1 patient of 6.

Secondary objectives are:

• Study of pharmacokinetics (PK) of multiple dosing of Quisinostat administered in combination with chemotherapy, as follows: Gemcitabine + Cisplatin in patients with non-small-cell lung cancer (second line) and Paclitaxel + Carboplatin in patients with non-small-cell lung cancer (second line) and in patients with ovarian cancer (second and subsequent lines) Preliminary estimation of possible effect of the drug, added to chemotherapy, on tumor growth.

ELIGIBILITY:
Inclusion Criteria:

General criteria for the inclusion of patients with non-small cell lung cancer (NSCLC) and ovarian cancer (OC):

1. Signed patient's information sheet and informed consent form to participate in the study
2. Age 18 and older
3. The value of left ventricular ejection fraction, as determined by echocardiography data, more than 50%
4. Patient's ability to carry out visits and study procedures and to comply with the protocol
5. Requirements to laboratory parameters determined below:

   Complete blood count: Absolute neutrophil count:

   Platelets:

   Haemoglobin: ≥ 1500/mm3 (1.5 x 109 cells/l)
   * 100 000/mm3 (100 x 109 cells/l)
   * 9.0 g/dl

   Liver function: Total bilirubin:

   aspartate aminotransferase (AST) and alanine aminotransferase (ALT): ≤ 1.5-fold of the upper limit of normal (ULN)

   ≤ 2.5--fold of ULN or ≤ 5.0-fold of ULN in case of metastases in liver Kidney function: GRF (by Cockcroft-Gault equation) > 50 ml/min
6. The expected survival time not less than 6 months
7. Women and men of childbearing potential (not sterile or in menopause less than 2 years) must be practicing an effective method of birth control starting from the screening period, during the study and 6 months after the last administration of the investigational product. Effective methods include use a condom or diaphragm (barrier method) with spermicide.
8. Functional status of the patient according to the ECOG 0 - 2 Special criteria for patients with NSCLC
9. Histologically or cytologically confirmed diagnosis of non-resectable non-small-cell lung cancer
10. The progression of lung cancer after a maximum of one line of systemic anticancer therapy (adjuvant chemotherapy will be considered first-line therapy if the time from the moment of its completion until disease progression was less than 6 months)
11. No history of treatment with Gemcitabine if the patient is planned for inclusion in the group of chemotherapy with Cisplatin and Gemcitabine, or Paclitaxel if the patient is planned for inclusion in the group of Carboplatin and Paclitaxel.
12. Vital capacity of lung by spirometry data is more than 50% of normal at screening

    Special inclusion criteria for patients with ovarian cancer
13. Histologically confirmed diagnosis of ovarian cancer.
14. Progression after no more than three modes of anticancer drug therapy for ovarian cancer.

Exclusion Criteria:

1. Indications for X-ray therapy or chemoradiation therapy at the time of inclusion, regardless of the treated area;
2. Presence of clinical and/or radiological signs of metastases in the brain and meningeal structures (CNS);
3. Previous therapy with HDAC inhibitors
4. Any contraindications to the chemotherapy with Gemcitabine + Cisplatin or Paclitaxel + Carboplatin (in patients with lung cancer); contraindications to chemotherapy according to the standard chemotherapy combination scheme Paclitaxel + Carboplatin (in female patients with ovarian cancer);
5. Any contraindications to administration of glucocorticosteroids, antihistamine drugs, serotonin 5-HT3 receptor antagonists, aprepitant;
6. Any contraindications to forced rehydration and/or administration of forced diuresis (in case of lung cancer);
7. Conditions that require continuous use of oral anticoagulants, or clinically significant changes in blood coagulation parameters at screening (INR > 1.5, aPTT> 1.5 х ULN)
8. Conditions that require admission of prohibited drugs, or impossibility to replace those with allowed drugs in the study
9. Current infection or other systemic conditions constituting a contraindication to the intended chemotherapy;
10. Diseases of the digestive system which may infringe absorption of the investigational product (Crohn's disease, nonspecific ulcerative colitis, irritable bowel syndrome)
11. Clinically significant cardiovascular diseases including:

    * Myocardial infarction within 12 months before screening
    * Unstable angina within 12 months before screening
    * Congestive heart failure Class III or IV according to the New York Heart Association criteria (NYHA)
    * Clinically significant ventricular arrhythmia including ventricular tachycardia, ventricular fibrillation, history of cardiac arrest, atrioventricular block (Mobitz II or III), use of cardiostimulator
    * QTc interval > 450 ms in men or 470 ms in women (ECG) (calculated according to Fredericia formula), or a diagnosis of long QT syndrome
    * Hypotension (systolic blood pressure < 86 mm Hg or bradycardia with a heart rate of < 50 beats per minute (ECG) except when caused by medications (e.g. beta-blockers).
    * Uncontrolled arterial hypertension (systolic arterial pressure > 170 millimeters of mercury or diastolic blood pressure > 105 millimeters of mercury)
12. Pregnancy and lactation
13. Presence of HIV antibodies, Hepatitis В and С antibodies
14. Drug or alcohol abuse at the moment of screening or in the past which according to the opinion of the Investigator makes the patient unsuitable for participation in the study
15. Significant allergic reactions in medical history
16. Participation in other clinical studies or administration of test drugs during 30 days before beginning of the study or persisting side effect of any of the test drugs;
17. Toxic effects of previous treatments or complications after surgical treatments that did not resolve to grades 1 and/or 0 (according to the CTCAE scale).
18. Patient not willing to participate in the study or unable to understand or follow the protocol instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of Quisinostat based on number of patients with treatment -related AEs assessed by CTCAE v4.0, number of patients with abnormal laboratory values and instrumental tests (ECG) that are related to treatment | 22 weeks

OTHER OUTCOMES:
Peak Plasma Concentration (Cmax) of Quisinostat | Day 1, Day 7
Area under the Quisinostat plasma concentration versus time curve (AUC) | Day 1, Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Tjulandin, Prof, Principal Investigator — Russian Oncological Research Center n.a. N. N. Blokhin RAMS
Locations (6):
- Russia (6):
  - Russian Oncological Research Center n.a. N. N. Blokhin RAMS, Moscow
  - State Budgetary Healthcare Institution of Stavropol Territory "Pyatigorsk oncology dispensary", Pyatigorsk
  - Saint-Peterburg State Budgetary healthcare Institution "City Clinical Oncology Dispensary", Saint Petersburg
  - BioEq LLC, Saint Petersburg
  - State Budget Institution of healthcare "Saint-Petersburg clinical research and practical centre of specialized medical aid (oncology)", Saint Petersburg
  - State Healthcare Institution of Yaroslavl region "Regional Clinical oncology hospital", Yaroslavl

IPD SHARING:
Plan to Share IPD: No
Final results will be published